CLINICAL TRIAL: NCT02066220
Title: AN INTERNATIONAL PROSPECTIVE TRIAL ON MEDULLOBLASTOMA (MB) IN CHILDREN OLDER THAN 3 TO 5 YEARS WITH WNT BIOLOGICAL PROFILE (PNET 5 MB - LR and PNET 5 MB - WNT-HR), AVERAGE-RISK BIOLOGICAL PROFILE (PNET 5 MB -SR), OR TP53 MUTATION, AND REGISTRY FOR MB OCCURRING IN THE CONTEXT OF GENETIC PREDISPOSITION
Brief Title: International Society of Paediatric Oncology (SIOP) PNET 5 Medulloblastoma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsche Kinderkrebsstiftung (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIOP PNET 5 MB; 2011-004868-30 (EudraCT Number)
Record Dates: First submitted 2014-02-07; First posted 2014-02-19 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumors
Keywords: pediatric brain tumor; medulloblastoma; event-free survival (EFS); progression-free survival (PFS); overall survival (OS); PNET; posterior fossa; chemotherapy; radiotherapy; biological profile; ß-catenin
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma; Neuroectodermal Tumors, Primitive | interventions — Radiotherapy; Carboplatin; Cisplatin; Lomustine; Vincristine; Cyclophosphamide; Maintenance Chemotherapy; Induction Chemotherapy; Diploidy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PNET 5 MB-LR (low-risk) (Experimental): Radiotherapy and reduced-intensity maintenance chemotherapy. Total treatment duration is 39 weeks.
  Interventions: Radiation: Radiotherapy without Carboplatin; Drug: Reduced-intensity maintenance chemotherapy
- PNET 5 MB-SR (standard-risk) (Experimental): Radiotherapy with carboplatin or radiotherapy without carboplatin and maintenance chemotherapy.
  Total treatment duration is 48 weeks.
  Interventions: Radiation: Radiotherapy without Carboplatin; Radiation: Radiotherapy with Carboplatin; Drug: Maintenance chemotherapy
- PNET 5 MB WNT-HR (Experimental): Radiotherapy adapted to age and metastatic Status and maintenance chemotherapy adapted to age.
  Total treatment duration is 39 to 48 weeks.
  Interventions: Drug: Maintenance chemotherapy; Radiation: WNT-HR < 16 years; Radiation: WNT-HR >= 16 years
- PNET 5 MB SHH-TP53 (Experimental): Reduced chemotherapy with Doxorubicin, VCR, HD-MTX, Carboplatin, and MTX intraventricularly Stratification of radiotherapy according to
  * presence of metastasis
  * germline mutation in TP53 (including mosaicism) Maintenance chemotherapy with VBL Total treatment duration is 1 year
  Interventions: Drug: Induction Chemotherapy; Radiation: SHH-TP53 M0; Radiation: SHH-TP53 M+ (germline); Radiation: SHH-TP53 (somatic); Drug: Vinblastin Maintenance

INTERVENTIONS:
Radiation: Radiotherapy without Carboplatin — Brain - 23.40 Gy in 13 daily fractions of 1.80 Gy Spine - 23.40 Gy in 13 daily fractions of 1.80 Gy Primary tumour boost - 30.60 Gy in 17 daily fractions of 1.80 Gy Total dose - 54 Gy Duration of radiotherapy 6 weeks
  LR Arm after Amendment (Protocol version 11- 17 Nov 2014):
  Brain - 18.0 Gy in 10 daily fractions of 1.80 Gy Spine - 18.0 Gy in 10 daily fractions of 1.80 Gy Primary tumour boost - 36.0 Gy in 20 daily fractions of 1.80 Gy Total dose - 54 Gy Duration of radiotherapy 6 weeks
  Arms: PNET 5 MB-LR (low-risk); PNET 5 MB-SR (standard-risk)
Drug: Reduced-intensity maintenance chemotherapy — Starts 6 weeks after radiotherapy. 6 cycles alternating Regimen A and Regimen B. Regimen A (cycles 1, 3, 5): cisplatin 70 mg/m2 day 1, CCNU 75 mg/m2 day 1, vincristine 1.5 mg/m2 days 1, 8 and 15, Regimen B: (cycles 2, 4, 6): cyclophosphamide 1 x 1000 mg/m2 days 1-2, vincristine 1.5 mg/m2 day 1.
  Interval after cycle A: 6 weeks, after cycle B: 3 weeks, for a total duration of 27 weeks.
  Cumulative doses of chemotherapy drugs: cisplatin 210 mg/m2, lomustine (CCNU) 225 mg/m2, vincristine 18 mg/m2, cyclophosphamide 6 g/m2.
  Other Names: Cisplatin; Lomustin (CCNU); Vincristine; Cyclophosphamide
  Arms: PNET 5 MB-LR (low-risk)
Radiation: Radiotherapy with Carboplatin — Brain - 23.40 Gy in 13 daily fractions of 1.80 Gy Spine - 23.40 Gy in 13 daily fractions of 1.80 Gy Primary tumour boost - 30.60 Gy in 17 daily fractions of 1.80 Gy Total dose - 54 G Carboplatin 35 mg/m2 5 times/week.
  Other Names: Carboplatin
  Arms: PNET 5 MB-SR (standard-risk)
Drug: Maintenance chemotherapy — Starts 6 weeks after radiotherapy. 8 cycles alternating Regimen A and Regimen B. Regimen A (cycles 1, 3, 5, 7): cisplatin 70 mg/m2 day 1, CCNU 75 mg/m2 day 1, vincristine 1.5 mg/m2 days 1, 8 and 15 Regimen B: (cycles 2, 4, 6, 8): cyclophosphamide 1 x 1000 mg/m2 days 1-2, vincristine 1.5 mg/m2 day 1.
  Interval after cycle A: 6 weeks, after cycle B: 3 weeks. Duration 36 weeks. Cumulative doses of chemotherapy drugs: cisplatin 280 mg/m2, lomustine (CCNU) 300 mg/m2, vincristine 24 mg/m2, cyclophosphamide 8 g/m2, carboplatin 1050 mg/m2 (in randomized patients).
  Other Names: Cisplatin; Lomustine (CCNU); Vincristine; Cyclophosphamide
  Arms: PNET 5 MB WNT-HR; PNET 5 MB-SR (standard-risk)
Radiation: WNT-HR < 16 years — Brain - 23.4 Gy in 13 daily fractions of 1.8 Gy Spine - 23.4 Gy in 13 daily fractions of 1.8 Gy Primary tumour boost - 30.6 Gy in 17 daily fractions of 1.8 Gy Boost to macroscopic metastases - 21.6 Gy in 12 daily fractions of 1.8 Gy Total dose to primary tumour - 54.0 Gy in 30 daily fractions of 1.8 Gy Total dose to cranial metastases - 45.0 Gy in 25 daily fractions of 1.8 Gy Total dose to spinal metastases - 45.0 Gy in 25 daily fractions of 1.8 Gy
  Arms: PNET 5 MB WNT-HR
Radiation: WNT-HR >= 16 years — Brain - 36.0 Gy in 20 daily fractions of 1.8 Gy Spine - 36.0 Gy in 20 daily fractions of 1.8 Gy Primary tumour boost - 18.0 Gy in 10 daily fractions of 1.8 Gy Metastases boost (cranial) - 14.4 Gy in 8 daily fractions of 1.8 Gy Metastases boost (spinal) - 9.0 Gy in 5 daily fractions of 1.8 Gy Total dose to primary tumour - 54.0 Gy in 30 daily fractions of 1.8 Gy Total dose to cranial metastases - 50.4 Gy in 30 daily fractions of 1.8 Gy Total dose to spinal metastases - 45.0 Gy in 25 daily fractions of 1.8 Gy
  Arms: PNET 5 MB WNT-HR
Drug: Induction Chemotherapy — Doxorubicin 37,5mg/m² in 24h-infusion, days 1 and 2 (If administration of doxorubicin is not deemed appropriate, doxorubicin can be substituted by carboplatin 200mg/m²) VCR 1,5mg/m² (max. dose 2mg) in short infusion, days 1, 15, 29, 43 HD-MTX 5g/m²in two doses (0.5g/m² in 0.5h and 4.5g/m² in 23.5h), days 15 and 29 (+ Leucovorin) Carboplatin 200mg/m² in 1h-infusion, days 43, 44, and 45 MTX 2mg intraventricularly, days 1-4, 15, 16, 29, 30, 43-46
  Arms: PNET 5 MB SHH-TP53
Radiation: SHH-TP53 M0 — * with VCR 1,5 mg/m2 (max. 2mg), once weekly during radiotherapy, for a maximum of 6 weeks
  * clinical target volume (CTV): safety margin along typical spread 10 mm: 23.4.Gy in 13 fractions to CTV.
  * focal RT boost to tumour bed and residual tumour (GTV) (boost: 30.6 Gy in 17 daily fractions of 1.8 Gy)
  Arms: PNET 5 MB SHH-TP53
Radiation: SHH-TP53 M+ (germline) — craniospinal radiotherapy with boost to tumour bed, residual tumour and metastatic deposits with VCR 1,5 mg/m2 (max. 2mg), once weekly during radiotherapy, for a maximum of 6 weeks Brain - 23.4 Gy in 13 daily fractions of 1.8 Gy Spine - 23.4 Gy in 13 daily fractions of 1.8 Gy Primary tumour boost - 30.6 Gy in 17 daily fractions of 1.8 Gy Metastases boost (cranial) - 30.6 Gy in 17 daily fractions of 1.8 Gy Metastases boost (spinal) - 21.6 Gy in 12 daily fractions of 1.8 Gy Total dose to primary tumour - 54.0 Gy in 30 daily fractions of 1.8 Gy Total dose to cranial metastases - 54.0 Gy in 30 daily fractions of 1.8 Gy Total dose to spinal metastases - 45.0 Gy in 25 daily fractions of 1.8 Gy
  Arms: PNET 5 MB SHH-TP53
Radiation: SHH-TP53 (somatic) — craniospinal radiotherapy with boost to tumour bed, residual tumour and metastatic deposits with VCR 1,5 mg/m2 (max. 2mg), once weekly during radiotherapy, for a maximum of 6 weeks Brain - 36.0 Gy in 20 daily fractions of 1.8 Gy Spine - 36.0 Gy in 20 daily fractions of 1.8 Gy Primary tumour boost - 18.0 Gy in 10 daily fractions of 1.8 Gy Metastases boost (cranial) - 18.0 Gy in 10 daily fractions of 1.8 Gy Metastases boost (spinal) - 9.0 Gy in 5 daily fractions of 1.8 Gy Total dose to primary tumour - 54.0 Gy in 30 daily fractions of 1.8 Gy Total dose to cranial metastases - 54.0 Gy in 30 daily fractions of 1.8 Gy Total dose to spinal metastases - 45 Gy in 25 daily fractions of 1.80 Gy
  Arms: PNET 5 MB SHH-TP53
Drug: Vinblastin Maintenance — Weekly VBL (5mg/m², max. 10mg/dose) for 24 weeks
  Arms: PNET 5 MB SHH-TP53

SUMMARY:
The study PNET 5 MB has been designed for children with medulloblastoma of standard risk (according to the risk-group definitions which have been used so far; e.g. in PNET 4). With the advent of biological parameters for stratification into clinical medulloblastoma trials, the ß-catenin status will be the only criterion according to which study patients will be assigned to either treatment arm PNET 5 MB - LR or to PNET 5 MB - SR, respectively. The initial diagnostic assessments (imaging, staging, histology, and tumor biology) required for study entry are the same for both treatment arms. With the amendment for version 12 of the protocol, patients who have a WNT-activated medulloblastoma with clinically high-risk features can be included in the PNET 5 MB WNT-HR study, and patients with a high-risk SHH medulloblastoma with TP53 mutation (both somatic or germline including mosaicism) can be included in the PNET5 MB SHH-TP53 study.

Data on patients with pathogenic germline alteration or cancer predisposition syndrome, who cannot be included in any prospective trial due to unavailability or due to physician or family decision, can be documented within the observational PNET 5 MB registry.

DETAILED DESCRIPTION:
The aim of the LR-study is to confirm the high rate of event-free survival in patients between the ages of 3 to 5 years and less than 22, with 'standard risk' medulloblastoma with a low-risk biological profile. Patients eligible for the study will be those with non-metastatic medulloblastoma (by CSF cytology and centrally reviewed MRI imaging) at diagnosis and low-risk biological profile, defined as ß-catenin nuclear immuno-positivity by immuno-histochemistry (IHC). Patients will have undergone total or near-total tumour resection and will receive conventionally fractionated (once a day) radiotherapy with a dose of 54 Gy to the primary tumor and 18.0 Gy to the craniospinal axis. Following radiotherapy, patients will receive a reduced-intensity chemotherapy with a total of 6 cycles of chemotherapy consisting of 3 courses of cisplatin, CCNU and vincristine alternating with 3 courses of cyclophosphamide and vincristine.

The aim of the SR-study is to test whether concurrent carboplatin during radiotherapy followed by 8 cycles of maintenance chemotherapy in patients with 'standard risk' medulloblastoma with an average-risk biological profile may improve outcome. Patients eligible for the study will be those with non-metastatic medulloblastoma (by CSF cytology and centrally reviewed MRI imaging) at diagnosis and average-risk biological profile, defined as ß-catenin nuclear immuno-negativity by IHC. Patients will have undergone total or near-total tumour resection and will receive conventionally fractionated (once a day) radiotherapy with a dose of 54 Gy to the primary tumor and 23.4 Gy to the craniospinal axis. Following radiotherapy, patients will receive a modified-intensity chemotherapy with a total of 8 cycles of chemotherapy consisting of 4 courses of cisplatin, CCNU and vincristine alternating with 4 courses of cyclophosphamide and vincristine.

The primary aim of the WNT-HR study is to maintain a 3-year EFS over 80 %. The small number of patients does not allow neither conventional methods of test size and power, nor strict stopping rules. The 3-year EFS will be estimated by the Kaplan-Meier method at the end of the trial and its two-sided 95 % confidence interval will be calculated.

The primary endpoint of the SHH-TP53 study is event-free survival (EFS). The aim of the study is the comparison of EFS between patients receiving a dose reduced induction chemotherapy, radiotherapy and maintenance chemotherapy and a historic population from unpublished data.

ELIGIBILITY:
Inclusion Criteria:

1. Age at diagnosis, at least 3 - 5 years (depending on the country) and less than 22 years (LR-arm: less than 16 years). The date of diagnosis is the date on which surgery is undertaken.
2. Histologically proven medulloblastoma, including the following subtypes, as defined in the WHO classification (2007): classic medulloblastoma, desmoplastic/nodular medulloblastoma. Pre-treatment central pathology review is considered mandatory.
3. Standard-risk medulloblastoma, defined as;

   * total or near total surgical resection with less than or equal to 1.5 cm2 (measured on axial plane) of residual tumour on early post-operative MRI, without and with contrast, on central review;
   * no central nervous system (CNS) metastasis on MRI (cranial and spinal) on central review;
   * no tumour cells on the cytospin of lumbar CSF
   * no clinical evidence of extra-CNS metastasis; Patients with a reduction of postoperative residual tumor through second surgery to less than or equal to 1.5 cm2 are eligible, if if timeline for start of radiotherapy can be kept.
4. Submission of high quality biological material including fresh frozen tumor samples for the molecular assessment of biological markers (such as the assessment of myelocytomatosis oncogene (MYC) copy number status) in national biological reference centers. Submission of blood is mandatory for all patients, who agree on germline DNA studies. Submission of CSF is recommended.
5. No amplification of MYC or MYCN (determined by FISH).
6. For LR-arm: Low-risk biological profile, defined as WNT subgroup positivity. The WNT subgroup is defined by the presence of (i) ß-catenin mutation (mandatory testing), or (ii) ß-catenin nuclear immuno-positivity by IHC (mandatory testing) and ß-catenin mutation, or (iii) ß-catenin nuclear immuno-positivity by IHC and monosomy 6 (optional testing).

   For SR-arm: average-risk biological profile, defined as ß-catenin nuclear immuno-negativity by IHC (mandatory) and mutation analysis (optional).
7. No prior therapy for medulloblastoma other than surgery.
8. Radiotherapy aiming to start no more than 28 days after surgery. Foreseeable inability to start radiotherapy within 40 days after surgery renders patients ineligible for the study.
9. Screening for the compliance with eligibility criteria should be completed, and patient should be included into the study within 28 days after first surgery (in case of second surgery within 35 days after first surgery). Inclusion of patients is not possible later than 40 days after first tumour surgery, or after start of radiotherapy.
10. Common toxicity criteria (CTC) grades < 2 for liver, renal, haematological function
11. no significant sensorineural hearing deficit as defined by pure tone audiometry with bone conduction or air conduction and normal tympanogram showing no impairment ≥ 20 decibel (dB) at 1-3 kilohertz (kHz). If performance of pure tone audiometry is not possible postoperatively, normal otoacoustic emissions are acceptable, if there is no history for hearing deficit.
12. No medical contraindication to radiotherapy or chemotherapy, such as preexisting DNA breakage syndromes (e.g. Fanconi Anemia, Nijmegen breakage syndrome), Gorlin Syndrome or other reasons as defined by patient's clinician.
13. No identified Turcot and Li Fraumeni syndrome.
14. Written informed consent (and patient assent where appropriate) for therapy according to the laws of each participating country. Information must be provided to the patient on biological studies (tumour and germline), and written informed consent obtained of agreement for participation.
15. National and local ethical committee approval according to the laws of each participating country (to include approval for biological studies).

Exclusion Criteria:

1. One of the inclusion criteria is lacking.
2. Brainstem or supratentorial primitive neuro-ectodermal tumour.
3. Atypical teratoid rhabdoid tumour.
4. Medulloepithelioma; Ependymoblastoma
5. Large-cell medulloblastoma, anaplastic medulloblastoma, or medulloblastoma with extensive nodularity (MBEN), centrally confirmed.
6. Unfavourable or undeterminable biological profile, defined as amplification of MYC or MYCN, or MYC or MYCN or WNT subgroup status not determinable.
7. Metastatic medulloblastoma (on CNS MRI and/or positive cytospin of postoperative lumbar CSF).
8. Patient previously treated for a brain tumour or any type of malignant disease.
9. DNA breakage syndromes (e.g. Fanconi anemia, Nijmegen breakage syndrome) or other, or identified Gorlin,Turcot, or Li Fraumeni syndrome.
10. Patients who are pregnant.
11. Female patients who are sexually active and not taking reliable contraception.
12. Patients who cannot be regularly followed up due to psychological, social, familial or geographic reasons.
13. Patients in whom non-compliance with toxicity management guidelines can be expected.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2014-06; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
3-year Event-Free Survival (EFS) | LR-arm after 9 years, SR-arm after 105 events (approx. 10 years)

SECONDARY OUTCOMES:
Overall survival | 10 years
Pattern of relapse | 10 years
  Defined in 5 categorical variables:
  no relapse, local relapse, distant relapse, local and distant relapse, death
Late effects of therapy on endocrine function | 10 years
  measured as
  1. subfertility (FSH > 15 IU/L)
  2. endocrine deficits (hormone supplementation necessary)
  3. growth retardation (calculated as the difference in height standard deviation score from diagnose) 2 and 5 years after diagnosis and age of 18 years
Late effects of therapy on audiology | 8 years
  measured on audiogram performed 2 years after diagnosis, grading according to Chang ototoxicity grading (Chang and Chinosornvatana 2010)
Late effects of therapy on neurology | 10 years
  Measured as
  1. presence, duration, and therapy of hydrocephalus symptoms (pre- and post-operatively)
  2. presence of posterior fossa syndrome (cerebellar mutism survey after surgery, before radiotherapy)
  3. cerebellar symptoms (brief ataxia rating scales 2 and 5 years after diagnosis and age of 18 years)
  4. presence of symptoms for brain nerve dysfunction (2 and 5 years after diagnosis and age of 18 years)
Late effects of therapy on quality of survival | 10 years
  measured with standardized questionnaires/ scores:
  1. HUI3 (health status)
  2. BRIEF (executive functions)
  3. SDQ (behavioural outcome)
  4. PedsQL (quality of life)
  5. QLQ-C30 (quality of life)
  6. MEES (neurological function, educational provision)
  7. MFI (fatigue) 2 and 5 years after diagnosis and age of 18 years
Progression-free survival | 10 years
Feasibility of carboplatin treatment | approx. 7 years
  measured as timely delivery of chemotherapy number of interruptions days during radiotherapy toxicities within 8 weeks after end of radiotherapy
Residual tumor | 6 years
  measured by central MRI review postoperatively
Leukoencephalopathy grading | 8 years
  measured 2 years after diagnosis grades 0, 1, 2, 3, 4

CONTACTS AND LOCATIONS:
Overall Officials: Francois Doz, Prof. Dr., Principal Investigator — Institut Curie Paris, France; Till Milde, Dr. med., Principal Investigator — Hopp Children´s Tumor Center at the NCT (KiTZ) and German Cancer Research Center
Locations (77):
- Medical University of Graz, Graz, Austria
- University Hospital Gasthuisberg, Leuven, Belgium
- University Hospital Brno, Brno, Czechia
- Rigshospitalet, Copenhagen, Denmark
- France (4):
  - CHU de Grenoble, Grenoble
  - Institute Curie, Paris
  - CHU-TOURS - Hôpital Clocheville, Tours
  - Hôpital NANCY-BRABOIS, Vandœuvre-lès-Nancy
- Germany (59):
  - University Hospital Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Helios Klinikum Berlin-Buch, Berlin
  - Charite Campus, University of Berlin, Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - University Hospital Bonn, Bonn
  - Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Chemnitz, Chemnitz
  - Kliniken der Stadt Köln, Cologne
  - University Hospital Cologne, Cologne
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Vestische Kinder- und Jugendklinik, University Witten/Herdecke, Datteln
  - Klinikum Dortmund, Dortmund
  - University Hospital Dresden, Dresden
  - Klinikum Duisburg, Duisburg
  - University Hospital Düsseldorf, Düsseldorf
  - HELIOS Klinikum-Erfurt, Erfurt
  - University Hospital Erlangen, Erlangen
  - University Hospital Essen, Essen
  - University Hospital Frankfurt/Main, Frankfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Gießen and Marburg, Giessen
  - University Hospital Göttingen, Göttingen
  - University Hospital Greifswald, Greifswald
  - University Hospital Halle/Saale, Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Angelika-Lautenschläger-Klinik, Heidelberg
  - Gemeinschaftskrankenhaus Herdecke, Herdecke
  - University Hospital Homburg/Saar, Homburg
  - University Hospital Jena, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikum Kassel, Kassel
  - UK-SH Campus Kiel, Kiel
  - Gemeinschaftsklinikum Koblenz-Mayen, Koblenz
  - HELIOS Klinikum Krefeld, Krefeld
  - University Hospital Leipzig, Leipzig
  - University Hospital Lübeck, Lübeck
  - University Hospital Magdeburg, Magdeburg
  - University Hospital Mainz, Mainz
  - University Hospital Mannheim, Mannheim
  - Johannes Wesling Klinikum Minden, Minden
  - University Hospital München, Dr. von Haunersches Kinderspital, München
  - Klinikum Schwabing, Pediatric Hospital of Technical University, München
  - University Hospital Münster, Münster
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - University Hospital Regensburg, Regensburg
  - University Hospital Rostock, Rostock
  - Asklepios Klinik Sankt Augustin, Sankt Augustin
  - HELIOS-Kliniken Schwerin, Schwerin
  - Klinikum Stuttgart, Stuttgart
  - Mutterhaus der Borromäerinnen, Trier
  - University Hospital Tübingen, Tübingen
  - University Hospital Ulm, Ulm
  - Dr. Horst Schmidt Kliniken, Wiesbaden
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - University Hospital Würzburg, Würzburg
- Our Lady's Children's Hospital, Dublin, Ireland
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy
- Prinses Máxima Center for Pediatric Oncology, Bilthoven, Netherlands
- Rigshospitalet, Oslo, Norway
- The Children's Memorial Health Institute, Warsaw, Poland
- University Hospital S.Joao, Porto, Portugal
- Oncology Hospital Cruces Bilbao, Barakaldo, Spain
- Barncancercentrum Drottning Silvias Barnochungdomssjukhus, Göteburg, Sweden
- University Children's Hospital, Zurich, Switzerland
- Great Ormond Street Hospital, London, United Kingdom